CLINICAL TRIAL: NCT03279315
Title: Exploration of the Appropriate Recommended Nutrient Intake of Iodine in Chinese Euthyroid Women: an Iodine Balance Experiment
Brief Title: An Iodine Balance Experiment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Wanqi Zhang, Professor, Tianjin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NSFC-31340033
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Iodine Deficiency; Nutritional Requirements
Keywords: Iodine; Balance experiment; EAR; Chinese women; Euthyroid

STUDY DESIGN:
Intervention Model Description: Participants received a diet with iodized table salt or non-iodized table salt
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental period (Experimental): the first period was with non-iodized salt, the second period was with iodized salt.
  Interventions: Dietary Supplement: iodized table salt, non-iodized table salt

INTERVENTIONS:
Dietary Supplement: iodized table salt, non-iodized table salt — During the first 3 weeks, the diet was provided with non-iodized salt, while the diet with iodized salt was only offered in the last week.

SUMMARY:
A 4-week study was conducted in 25 Chinese euthyroid women. Unified diets with different iodine contents (cooked with non-iodized salt or iodized salt) were provided in two different periods. The total iodine intake from diet, water and air as well as the total iodine excretion by urine, faces and respiration were monitored and determined, and a total of 300 samples were collected. The sweat iodine loss was also considered. Moreover, the regression curve model between the 24-h iodine intake and 24-h iodine excretion was also established.

DETAILED DESCRIPTION:
The experiment was conducted between November and December with a total duration of 1 month. Referring to the experience from Harrison and Dworkin, however, considering the negative iodine balance reported, during the first 3 weeks, the diet was provided with non-iodized salt, while the diet with iodized salt was only offered in the last week. The total daily iodine intake consisted of dietary iodine intake, water iodine intake and iodine from breathing, while iodine could be excreted out of human body by urine, faces, sweat and breathing. The 24-h iodine intake and 24-h iodine excretion were determined in each individual participant, and the iodine balance was calculated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* The ones with normal thyroid function, urinary iodine concentration, agree with the experiment.

Exclusion Criteria:

* The ones with abnormal thyroid hormone level, urinary iodine concentration (UIC) or autoantibody-positive were excluded from the study.

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11-20 (Actual); Primary Completion 2014-12-19 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Total iodine intake and total iodine excretion | 12 days
  Iodine intake includes iodine from food, water and air (μg/d).
Total iodine excretion | 12 days
  Iodine excretion includes iodine excreted by urine, feces, sweat and breath (μg/d).
urinary iodine concentration (UIC) | At the beginning of the experiment
  μg/L
Thyroid function | At the beginning of the experiment
  FT3 (pmol/L), FT4 (pmol/L),TSH (mIU/L), TG (ng/mL), TGAb (IU/mL), TPOAb (IU/mL)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Tian X, Song Q, Wang W, Guo X, Cui T, Pan Z, Chen Y, Chen W, Tan L, Zhang W. Application and Comparison of Different Regression Models in Iodine Balance Experiment on Women of Childbearing Age and Pregnant Women. Biol Trace Elem Res. 2024 Jun;202(6):2474-2487. doi: 10.1007/s12011-023-03867-x. Epub 2023 Oct 9. PMID 37807000